CLINICAL TRIAL: NCT00381394
Title: A Phase II, Multi-centre, Open-label, Randomised Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Oral Sitamaquine Compared With Amphotericin B in the Treatment of Visceral Leishmaniasis Caused by L. Donovani in Endemic Areas.
Brief Title: A Study Evaluating Sitamaquine Compared With Amphotericin B In The Treatment Of Visceral Leishmaniasis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STQ105938
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Leishmaniasis, Visceral
Keywords: amphotericin B; safety; tolerability and pharmacokinetics of oral sitamaquine; Visceral leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — 8-aminoquinoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sitamaquine

SUMMARY:
Sitamaquine is an 8-aminoquinoline which is being developed as an oral treatment for visceral leishmaniasis (VL). Pre-clinical and subsequent clinical investigations have demonstrated oral efficacy against Leishmania donovani. The purposes of this study are to characterise the pharmacokinetic profile of sitamaquine, administered orally, and to determine if the pharmacokinetic profile is affected by administration with food. The study is also designed to further characterise the safety and tolerability of sitamaquine compared with amphotericin B, particularly in reference to renal, hepatic and cardiac adverse events, prior to initiation of phase III studies. Finally the study will investigate the efficacy of a 21 day treatment course. Previous studies have used 28 days dosing, but parasitological evidence from one study suggests that shorter courses may be effective.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of visceral leishmaniasis; symptoms and signs compatible with VL and diagnosis confirmed by visualisation of amastigotes in splenic aspirate or bone marrow.
* Written informed consent or witnessed oral consent.
* Willing to comply with the study visits and procedures.
* For female subjects, a negative urine pregnancy test at screening and before dosing and the subject agrees to use an established method of birth control (including abstinence).

Exclusion criteria:

* Past history of renal disease or impaired renal function at screening.
* History of any significant hepatic or biliary disease, or the following abnormal laboratory values at screening; hepatic dysfunction (AST or ALT 2.5 times upper limit of normal).
* Subjects with the following abnormal laboratory values; haemoglobin 6.5 g/dl, neutrophils <750/ mm3, platelets <50,000 / mm3, any clinically relevant abnormality identified on screening examination or clinical laboratories which would preclude the subject's safe participation in the study.
* History of cardiac disease, arrhythmias, conduction abnormalities or any clinically relevant abnormality identified on 12-lead ECG at screening.

Subjects suffering from a concomitant infection, blood disorder or any other serious underlying disease which would preclude evaluation of the subject's response to the study medication.

Methaemoglobin levels >5% at screening. G6PD deficiency.

* Positive HIV antibody, hepatitis B surface antigen or hepatitis C antibody at screening.
* Pregnant or nursing women; women of childbearing potential who are unwilling or unable to use an appropriate form of contraception, from prior to study medication administration until 2 weeks following the last dose of investigational product.
* Any contraindication to splenic aspirate (or bone marrow aspirate), including but not limited to PT prolonged >3 seconds longer than control or platelets <50,000 / mm3.
* Subjects with a known hypersensitivity reaction to 8-aminoquinolines (e.g. primaquine) or any of the investigational product excipients.
* Treatment with an established antileishmanial chemotherapeutic agent within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2006-08-04 (Actual); Primary Completion 2007-09-14 (Actual); Study Completion 2007-09-14 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve over the dosing interval AUC(0-tau) for sitamaquine | At Day 1, 10 and 21: immediately pre-dose, and at 1, 2, 3, 4, 6, 10, 16 hours post dose
  AUC is defined as the area under the concentration-time curve from 0 to last quantifiable concentration (AUC 0-tau). AUC is a measure of exposure. Blood samples for determination of plasma concentrations of sitamaquine was obtained at the following time points on days 1, 10 and 21: immediately pre-dose, and at 1, 2, 3, 4, 6, 10, 16 hours post dose. An additional sample was taken on Day 23 and Day 24 to approximate 48 hours and 72 hours post last dose on Day 21. Only those participants with data available at the specified time points were analyzed.
Maximum plasma concentration (Cmax) for sitamaquine | At Day 1, 10 and 21: immediately pre-dose, and at 1, 2, 3, 4, 6, 10, 16 hours post dose.
  Cmax was defined as the maximum concentration of sitamaquine. Blood samples for determination of plasma concentrations of sitamaquine was obtained at the following time points on days 1, 10 and 21: immediately pre-dose, and at 1, 2, 3, 4, 6, 10, 16 hours. An additional sample was taken on Day 23 and Day 24 to approximate 48 hours and 72 hours post last dose on Day 21.
Time to maximum observed plasma concentration (tmax) for sitamaquine | At Day 1, 10 and 21: immediately pre-dose, and at 1, 2, 3, 4, 6, 10, 16 hours post dose.
  Tmax is defined as the time to peak concentration from initiation of sitamaquine dosing. Blood samples for determination of plasma concentrations of sitamaquine was obtained at the following time points on days 1, 10 and 21: immediately pre-dose, and at 1, 2, 3, 4, 6, 10, 16 hours post dose. An additional sample was taken on Day 23 and Day 24 to approximate 48 hours and 72 hours post last dose on Day 21.
Accumulation ratio for sitamaquine | At Day 1, 10 and 21: immediately pre-dose, and at 1, 2, 3, 4, 6, 10, 16 hours post dose
  Point estimate was the ratio of adjusted geometric means between repeat dosing days (Day 21 or Day 10) and single dose day (Day 1). An evaluation on the accumulation rate was based upon the comparison of AUC(0-24) values after repeated dosing to the values from the first dose on day 1. Blood samples for determination of plasma concentrations of sitamaquine was obtained at the following time points on days 1, 10 and 21: immediately pre-dose, and at 1, 2, 3, 4, 6, 10, 16 hours post dose. An additional sample was taken on Day 23 and Day 24 to approximate 48 hours and 72 hours post last dose on Day 21. Individual observed accumulation ratios on Day 10 were calculated by dividing AUC (0-tau) on Day 10 by AUC (0-tau) on Day 1. A similar formula was applied to the accumulation ratio on Day 21.

SECONDARY OUTCOMES:
Number of participants with adverse events(AEs) and serious adverse events(SAEs) | Up to 180 days
  An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Data for on-treatment AEs have been reported,
Number of participants with abnormal 12-lead Electrocardiogram (ECG) values | At Day 22 for Sitamaquine and Day 31 for Amphotericin B
  Data for abnormal findings have been reported at Day 22 for Sitamaquine and Day 31 for Amphotericin B. All ECGs were collected in the supine position with the electrodes placed in the standard positions, 4 hours after dosing on drug administration days, and prior to blood collection or pulse rate measurement.
Number of participants with abnormal echocardiography results | Up to Day 22 and 49 (sitamaquine only) and Day 31 and 58 (amphotericin B only)
  2-D echocardiograms were performed at screening (all participants), Days 22 and 49 (sitamaquine only) and days 31 and 58 (amphotericin B only). All echocardiograms were obtained after the participant has rested in a semi-supine position for at least 10 minutes. All echocardiograms were stored electronically (e.g video home system [VHS] tape, optical drive, etc.). Ejection fraction was estimated using the modified Simpson's rule method. Data for number of participants with abnormal echocardiography results have been reported.
Change from Baseline in systolic blood pressure (SBP) and diastolic blood pressure (DBP) at Day 180 | Baseline (Day 1 pre-dose) and Day 180
  Blood pressure (SBP and DBP) was recorded after the participant had rested in a semi-supine position for at least 10 minutes. Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was Day 1 pre-dose.
Change from Baseline in heart rate | Baseline (Day 1 pre-dose) and Day 180
  Heart rate was recorded after the participant had rested in a semi-supine position for at least 10 minutes. Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was Day 1 pre-dose.
Change from Baseline in body temperature | Baseline (Day 1 pre-dose) and Day 180
  Body temperature was recorded after the participant had rested in a semi-supine position for at least 10 minutes. Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was Day 1 pre-dose.
Change from Baseline in body weight | Baseline (Day 1 pre-dose) and Day 49 for Sitamaquine and Day 58 for Amphotericin B
  Body weight was recorded after the participant had rested in a semi-supine position for at least 10 minutes. Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was Day 1 pre-dose.
Number of participants with abnormal hematology values at the end of study (Day 180) | Day 180
  Data for number of participants with hematology abnormalities for the end of study (Day 180) is presented. Hematology abnormalities were classified using Common Terminology Criteria for Adverse Events (CTCAE) v3.0 Grades and grade 3 ranges are as follows (selected): Hemoglobin (grams per liter [G/L])- <80 - 65; Total Neutrophils (gram international units per liter[GI/L])- <1.0 - 0.5 x 10^9/L; Platelet count(GI/L) <50.0- 25.0 x 10^9 /L; White Blood Cell (WBC) (GI/L)- <2.0 - 1.0 x 10^9 /L. Data only for categories with values have been presented.
Number of participants with abnormal clinical chemistry values at the end of study (Day 180) | Day 180
  Aspartate Amino Transferase (AST) ([international units per liter [IU/L])- >5.0 - 20.0 x upper limit of normal (ULN); Albumin(G/L)- <20 g/dL; Alkaline Phosphatase(IU/L)- >5.0 - 20.0 x ULN; Alanine Amino Transferase(IU/L)- >5.0 - 20.0 x ULN; Total Bilirubin( micromoles per liter [µMOL/L])- >3.0 - 10.0 x ULN; Urea(millimoles per liter [MMOL/L])- 5.1 - 10 x ULN; Cholesterol (MMOL/L) - >10.34 - 12.92; Creatine Kinase MB (microgram per liter[µ/L])->5 x ULN - 10 x ULN; Creatinine Clearance(milliliter per minute [mL/min])- <25% lower limit of normal (LLN); Creatinine(µMOL/L)- >3.0 - 6.0 x ULN; Gamma Glutamyl Transferase(IU/L)- >5.0 - 20.0 x ULN; Potassium(MMOL/L)- >6.0 - 7.0(high) and <3.0 - 2.5 (low); Sodium(MMOL/L)- >155 - 160; Sodium(MMOL/L)- <130 - 120; Triglycerides(MMOL/L)- >5.0 - 10.0 x ULN. Data only for categories with values have been presented.
Number of participants with Initial parasitological cure (28 days) | Up to 28 days
  Initial parasitological cure was defined as a parasite-negative splenic aspirate at completion of treatment or, if the leishmania index (a quantitative assessment of parasites in the splenic aspirate) was +1, a parasite-negative result at the repeat splenic aspirate 28 days later.
Number of participants with Final parasitological cure (6 months) | Up to 180 days
  Final clinical cure was defined as initial parasitological cure (initial parasitological cure was defined as a parasite-negative splenic aspirate at completion of treatment or, if the leishmania index [a quantitative assessment of parasites in the splenic aspirate] was +1, a parasite-negative result at the repeat splenic aspirate 28 days later) and no evidence of relapse at 6 months.
Terminal elimination half-life (t1/2) for sitamaquine | At Day 1, 10 and 21: immediately pre-dose, and at 1, 2, 3, 4, 6, 10, 16 hours post dose
  Half life is defined as the period of time required for the amount of drug in the body to be reduced by half. Blood samples for determination of plasma concentrations of sitamaquine was obtained at the following time points on days 1, 10 and 21: immediately pre-dose, and at 1, 2, 3, 4, 6, 10, 16 hours post dose. An additional sample was taken on Day 23 and Day 24 to approximate 48 hours and 72 hours post last dose on Day 21.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- India (2):
  - GSK Investigational Site, Muzaffarpur
  - GSK Investigational Site, Patna

REFERENCES:
- [Result] Sundar S, Sinha PK, Dixon SA, Buckley R, Miller AK, Mohamed K, Al-Banna M. Pharmacokinetics of oral sitamaquine taken with or without food and safety and efficacy for treatment of visceral leishmaniais: a randomized study in Bihar, India. Am J Trop Med Hyg. 2011 Jun;84(6):892-900. doi: 10.4269/ajtmh.2011.10-0409. PMID 21633025